CLINICAL TRIAL: NCT04898803
Title: How Effective Can a Simulator-Based Training Course For Beginners In Endoscopy Be Made?
Acronym: EFFEKTRA
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Olympus Deutschland GmbH (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Clinical Director, Department of Interdisciplinary Endoscopy, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV7217
Record Dates: First submitted 2021-01-25; First posted 2021-05-24 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Physicians Gastroscopy Training
Keywords: simulator training; gastroscopy training; physicians training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conventional gastroscopy training course: physicians receive the DGVS-recommended training, consisting of a 2-day course with 1 hour of simulator training
  Interventions: Other: conventional DGVS training
- extended simulator course: physicians receive a two-day simulator course with a minimum of 6 hours of simulator training per trainee, structured in stages in the sense of progressive or mastery learning. The initial part of the training will be part-task training.
  Interventions: Other: extended simulator training

INTERVENTIONS:
Other: conventional DGVS training — see above
  Groups: conventional gastroscopy training course
Other: extended simulator training — see above
  Groups: extended simulator course

SUMMARY:
The aim of the study is to clarify whether physicians training for gastroscopies benefit from a modified training course. The duration and type of optimized use of training simulators as part of a basic gastroscopy course can lead to a higher level of competence in patient examinations (main target parameters) than conventional use. Further goals are the comparison of the theoretical knowledge gained through the modified versus conventional course, as well as the self-assessment of the participants.

DETAILED DESCRIPTION:
Training in interventional medicine, including surgery and endoscopy, is usually still done on the patient, under more or less qualified supervision. Previous exercises on models or simulators are still the exception and only reach around 40% of colleagues in countries with defined curricula and guidelines.The simulator-based training, however, offers a protected area in which, without risk to the patient, initial learning successes in flexible endoscopy can be achieved according to the "trial and error" principle. Various studies have shown that initial training on the simulator is beneficial: Physicians trained on the simulator require less support during the first examinations on the patient, less examination time, can reach and identify anatomical landmarks better and have better hand-eye coordination.If the simulator training is embedded in a structured curriculum, greater successes seem to be achieved in comparison to unstructured training. The feedback during the training is also a positive influencing factor; this should ideally take place at the end of each unit. It is also possible to use a simulator to train defined partial performances and to repeat these in the required amount. A step-by-step structure with defined intermediate goals, in the sense of mastery learning, also increases effectiveness.There is little data on the optimal duration or the saturation of the learning curve in simulator training. In one study the learning curve flattened after 60 simulated colonoscopies. Another study showed a gradual improvement up to 6 hours on the simulator. It also used threshold values for the performance score to define the optimal point in time for transition to patient-based training.

The current certification for the standardization of the nationwide endoscopy training courses by the German Gastroenterological Society (DGVS), provides for 4 hours of training on the simulator, including one hour of introduction. With an also recommended maximum group size of 4 participants per simulator, this corresponds to a duration of only 1 hour of effective simulator training per trainee. There are no recommendations for structuring simulator trainings or the type of simulators used.

The main aim of the present study is to find out whether it is possible to improve this situation without unrealistically extending the training and course times.

Trainees will randomly attend either a conventional training or an extended simulator training. Immediately after the course, in accordance with the DGVS guidelines, an examination of the same content for both groups to inquire the theoretical knowledge is done.1-5 weeks after completion of the training course, an evaluation of the endoscopic skills of the participants takes place. It is done on the patient, under supervision, as is currently customary in everyday clinical training. After a one-day introduction through observation of routine gastroscopies, two gastroscopies are then carried out. Two endoscopists independently assess the performance based on a Video record of the examination. All endoscopists involved in supervision or assessment are blinded to the trainee's group membership..

ELIGIBILITY:
Inclusion Criteria:

Trainees:

* licensed physicians in internal medicine, surgery or gastroenterology,
* no endoscopic or laparoscopic experience
* informed consent

Patient's endoscopies:

* all patients > 18 years of age who are capable of being informed and have a clinical indication for esophagogastroduodenoscopy
* informed consent
* simple examination expected

Exclusion Criteria:

Patient's endoscopies:

- difficult examination expected

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: see above
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Global Assessment of Gastrointestinal Endoscopic Skills (GAGES) competence score competence score | one to five weeks after training course
  Comparison of the GAGES competence score of the video-based observations of the first two patient examinations, each assessed by two endoscopists. To be valuated: intubation of esophagus, scope navigation, ability to keep a clear endoscope field, instrumentation, quality of examination. Best score each question 5 pts, worst 1 pt.
Non-inferiority of the new training procedure | through study completion, approximately 1 year
  Non-inferiority of the new training procedure in the final exams according to DGVS criteria

SECONDARY OUTCOMES:
competence assessment Direct Observation of Procedural Skills (DOPS) by Joint Advisory Group on Gastrointestinal Endoscopy (JAG) | one to five weeks after training course
  Comparison of the JAG DOPS competence level of the video-based observations of the first two patient examinations, each assessed by two endoscopists. Assession of trainee's needed level of supervision at pre- and post procedure, insertion and withdrawal, visualisation, management of findings, and non-technical skills. Each has 4 values, best is "Competent for independent practice", worst is "maximal supervision"
Assessment of Competency in Endoscopy (ACE) | one to five weeks after training course
  Comparison of the ACE competence evaluation of the video-based observations of the first two patient examinations, each assessed by two endoscopists.
mean self-assessment by Visual Analog Scale (VAS) | one to five weeks after training course
  VAS after the first two patient examinations. This enables an assessment of the stress level and ultimately a measurement of the cognitive load of the subject. To be evaluated on a non-scaled line from "do not agree at all" to "totally agree".

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - University Hospital Eppendorf, Hamburg
  - Albertinen Krankenhaus, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amiot A, Conroy G, Le Baleur Y, Winkler J, Palazzo M, Treton X. Endoscopic training: A nationwide survey of French fellows in gastroenterology. Clin Res Hepatol Gastroenterol. 2018 Apr;42(2):160-167. doi: 10.1016/j.clinre.2017.08.005. Epub 2017 Sep 18. PMID 28927657
- [Background] Jirapinyo P, Thompson CC. Current status of endoscopic simulation in gastroenterology fellowship training programs. Surg Endosc. 2015 Jul;29(7):1913-9. doi: 10.1007/s00464-014-3884-0. Epub 2014 Oct 11. PMID 25303910
- [Background] Ende A, Zopf Y, Konturek P, Naegel A, Hahn EG, Matthes K, Maiss J. Strategies for training in diagnostic upper endoscopy: a prospective, randomized trial. Gastrointest Endosc. 2012 Feb;75(2):254-60. doi: 10.1016/j.gie.2011.07.063. Epub 2011 Dec 7. PMID 22153875
- [Background] Haycock A, Koch AD, Familiari P, van Delft F, Dekker E, Petruzziello L, Haringsma J, Thomas-Gibson S. Training and transfer of colonoscopy skills: a multinational, randomized, blinded, controlled trial of simulator versus bedside training. Gastrointest Endosc. 2010 Feb;71(2):298-307. doi: 10.1016/j.gie.2009.07.017. Epub 2009 Nov 3. PMID 19889408
- [Background] Sedlack RE, Kolars JC, Alexander JA. Computer simulation training enhances patient comfort during endoscopy. Clin Gastroenterol Hepatol. 2004 Apr;2(4):348-52. doi: 10.1016/s1542-3565(04)00067-9. PMID 15067632
- [Background] Shirai Y, Yoshida T, Shiraishi R, Okamoto T, Nakamura H, Harada T, Nishikawa J, Sakaida I. Prospective randomized study on the use of a computer-based endoscopic simulator for training in esophagogastroduodenoscopy. J Gastroenterol Hepatol. 2008 Jul;23(7 Pt 1):1046-50. doi: 10.1111/j.1440-1746.2008.05457.x. Epub 2008 Jun 28. PMID 18554236
- [Background] Ahlberg G, Hultcrantz R, Jaramillo E, Lindblom A, Arvidsson D. Virtual reality colonoscopy simulation: a compulsory practice for the future colonoscopist? Endoscopy. 2005 Dec;37(12):1198-204. doi: 10.1055/s-2005-921049. PMID 16329017
- [Background] Cohen J, Cohen SA, Vora KC, Xue X, Burdick JS, Bank S, Bini EJ, Bodenheimer H, Cerulli M, Gerdes H, Greenwald D, Gress F, Grosman I, Hawes R, Mullin G, Schnoll-Sussman F, Starpoli A, Stevens P, Tenner S, Villanueva G. Multicenter, randomized, controlled trial of virtual-reality simulator training in acquisition of competency in colonoscopy. Gastrointest Endosc. 2006 Sep;64(3):361-8. doi: 10.1016/j.gie.2005.11.062. PMID 16923483
- [Background] Di Giulio E, Fregonese D, Casetti T, Cestari R, Chilovi F, D'Ambra G, Di Matteo G, Ficano L, Delle Fave G. Training with a computer-based simulator achieves basic manual skills required for upper endoscopy: a randomized controlled trial. Gastrointest Endosc. 2004 Aug;60(2):196-200. doi: 10.1016/s0016-5107(04)01566-4. PMID 15278044
- [Background] Ferlitsch A, Schoefl R, Puespoek A, Miehsler W, Schoeniger-Hekele M, Hofer H, Gangl A, Homoncik M. Effect of virtual endoscopy simulator training on performance of upper gastrointestinal endoscopy in patients: a randomized controlled trial. Endoscopy. 2010 Dec;42(12):1049-56. doi: 10.1055/s-0030-1255818. Epub 2010 Oct 22. PMID 20972956
- [Background] Maiss J, Millermann L, Heinemann K, Naegel A, Peters A, Matthes K, Hahn EG, Hochberger J. The compactEASIE is a feasible training model for endoscopic novices: a prospective randomised trial. Dig Liver Dis. 2007 Jan;39(1):70-8; discussion 79-80. doi: 10.1016/j.dld.2006.07.007. Epub 2006 Aug 30. PMID 16942923
- [Background] McIntosh KS, Gregor JC, Khanna NV. Computer-based virtual reality colonoscopy simulation improves patient-based colonoscopy performance. Can J Gastroenterol Hepatol. 2014 Apr;28(4):203-6. doi: 10.1155/2014/804367. PMID 24729994
- [Background] Park J, MacRae H, Musselman LJ, Rossos P, Hamstra SJ, Wolman S, Reznick RK. Randomized controlled trial of virtual reality simulator training: transfer to live patients. Am J Surg. 2007 Aug;194(2):205-11. doi: 10.1016/j.amjsurg.2006.11.032. PMID 17618805
- [Background] Sedlack RE, Kolars JC. Computer simulator training enhances the competency of gastroenterology fellows at colonoscopy: results of a pilot study. Am J Gastroenterol. 2004 Jan;99(1):33-7. doi: 10.1111/j.1572-0241.2004.04007.x. PMID 14687137
- [Background] Tuggy ML. Virtual reality flexible sigmoidoscopy simulator training: impact on resident performance. J Am Board Fam Pract. 1998 Nov-Dec;11(6):426-33. doi: 10.3122/jabfm.11.6.426. PMID 9875997
- [Background] Yi SY, Ryu KH, Na YJ, Woo HS, Ahn W, Kim WS, Lee DY. Improvement of colonoscopy skills through simulation-based training. Stud Health Technol Inform. 2008;132:565-7. PMID 18391369
- [Background] Grover SC, Garg A, Scaffidi MA, Yu JJ, Plener IS, Yong E, Cino M, Grantcharov TP, Walsh CM. Impact of a simulation training curriculum on technical and nontechnical skills in colonoscopy: a randomized trial. Gastrointest Endosc. 2015 Dec;82(6):1072-9. doi: 10.1016/j.gie.2015.04.008. Epub 2015 May 23. PMID 26007221
- [Background] Grover SC, Scaffidi MA, Khan R, Garg A, Al-Mazroui A, Alomani T, Yu JJ, Plener IS, Al-Awamy M, Yong EL, Cino M, Ravindran NC, Zasowski M, Grantcharov TP, Walsh CM. Progressive learning in endoscopy simulation training improves clinical performance: a blinded randomized trial. Gastrointest Endosc. 2017 Nov;86(5):881-889. doi: 10.1016/j.gie.2017.03.1529. Epub 2017 Mar 31. PMID 28366440
- [Background] A Simulation-Based Training Curriculum of Progressive Fidelity and Complexity Improves Technical and Non-Technical Skills in Colonoscopy: a Blinded, Randomized Trial
- [Background] Harewood GC, Murray F, Winder S, Patchett S. Evaluation of formal feedback on endoscopic competence among trainees: the EFFECT trial. Ir J Med Sci. 2008 Sep;177(3):253-6. doi: 10.1007/s11845-008-0161-z. Epub 2008 Jun 27. PMID 18584274
- [Background] IMPACT OF A GAME-BASED LEARNING INTERVENTION IN SIMULATION-BASED ENDOSCOPY TRAINING ON COLONOSCOPY PERFORMANCE IN NOVICE ENDOSCOPISTS - A RANDOMIZED CONTROLLED TRIAL
- [Background] Hashimoto DA, Petrusa E, Phitayakorn R, Valle C, Casey B, Gee D. A proficiency-based virtual reality endoscopy curriculum improves performance on the fundamentals of endoscopic surgery examination. Surg Endosc. 2018 Mar;32(3):1397-1404. doi: 10.1007/s00464-017-5821-5. Epub 2017 Aug 15. PMID 28812161
- [Background] Ritter EM, Taylor ZA, Wolf KR, Franklin BR, Placek SB, Korndorffer JR Jr, Gardner AK. Simulation-based mastery learning for endoscopy using the endoscopy training system: a strategy to improve endoscopic skills and prepare for the fundamentals of endoscopic surgery (FES) manual skills exam. Surg Endosc. 2018 Jan;32(1):413-420. doi: 10.1007/s00464-017-5697-4. Epub 2017 Jul 11. PMID 28698900
- [Background] Hatala R, Cook DA, Zendejas B, Hamstra SJ, Brydges R. Feedback for simulation-based procedural skills training: a meta-analysis and critical narrative synthesis. Adv Health Sci Educ Theory Pract. 2014 May;19(2):251-72. doi: 10.1007/s10459-013-9462-8. Epub 2013 May 28. PMID 23712700
- [Background] Kruglikova I, Grantcharov TP, Drewes AM, Funch-Jensen P. The impact of constructive feedback on training in gastrointestinal endoscopy using high-fidelity Virtual-Reality simulation: a randomised controlled trial. Gut. 2010 Feb;59(2):181-5. doi: 10.1136/gut.2009.191825. Epub 2009 Oct 13. PMID 19828469
- [Background] Mahmood T, Darzi A. The learning curve for a colonoscopy simulator in the absence of any feedback: no feedback, no learning. Surg Endosc. 2004 Aug;18(8):1224-30. doi: 10.1007/s00464-003-9143-4. Epub 2004 Jun 23. PMID 15457382
- [Background] Vilmann AS, Norsk D, Svendsen MBS, Reinhold R, Svendsen LB, Park YS, Konge L. Computerized feedback during colonoscopy training leads to improved performance: a randomized trial. Gastrointest Endosc. 2018 Nov;88(5):869-876. doi: 10.1016/j.gie.2018.07.008. Epub 2018 Jul 19. PMID 30031803
- [Background] Walsh CM, Ling SC, Wang CS, Carnahan H. Concurrent versus terminal feedback: it may be better to wait. Acad Med. 2009 Oct;84(10 Suppl):S54-7. doi: 10.1097/ACM.0b013e3181b38daf. PMID 19907387
- [Background] Berger-Richardson D, Kurashima Y, von Renteln D, Kaneva P, Feldman LS, Fried GM, Vassiliou MC. Description and Preliminary Evaluation of a Low-Cost Simulator for Training and Evaluation of Flexible Endoscopic Skills. Surg Innov. 2016 Apr;23(2):183-8. doi: 10.1177/1553350615604054. Epub 2015 Sep 3. PMID 26337331
- [Background] Jirapinyo P, Abidi WM, Aihara H, Zaki T, Tsay C, Imaeda AB, Thompson CC. Preclinical endoscopic training using a part-task simulator: learning curve assessment and determination of threshold score for advancement to clinical endoscopy. Surg Endosc. 2017 Oct;31(10):4010-4015. doi: 10.1007/s00464-017-5436-x. Epub 2017 Feb 22. PMID 28229238
- [Background] Thompson CC, Jirapinyo P, Kumar N, Ou A, Camacho A, Lengyel B, Ryan MB. Development and initial validation of an endoscopic part-task training box. Endoscopy. 2014 Sep;46(9):735-44. doi: 10.1055/s-0034-1365463. Epub 2014 Apr 25. PMID 24770972
- [Background] Koch AD, Ekkelenkamp VE, Haringsma J, Schoon EJ, de Man RA, Kuipers EJ. Simulated colonoscopy training leads to improved performance during patient-based assessment. Gastrointest Endosc. 2015 Mar;81(3):630-6. doi: 10.1016/j.gie.2014.09.014. Epub 2014 Dec 2. PMID 25475901
- [Background] Vassiliou MC, Kaneva PA, Poulose BK, Dunkin BJ, Marks JM, Sadik R, Sroka G, Anvari M, Thaler K, Adrales GL, Hazey JW, Lightdale JR, Velanovich V, Swanstrom LL, Mellinger JD, Fried GM. Global Assessment of Gastrointestinal Endoscopic Skills (GAGES): a valid measurement tool for technical skills in flexible endoscopy. Surg Endosc. 2010 Aug;24(8):1834-41. doi: 10.1007/s00464-010-0882-8. Epub 2010 Jan 29. PMID 20112113
- [Background] Siau K, Crossley J, Dunckley P, Johnson G, Feeney M, Hawkes ND, Beales ILP; Joint Advisory Group on Gastrointestinal Endoscopy (JAG). Correction to: Direct observation of procedural skills (DOPS) assessment in diagnostic gastroscopy: nationwide evidence of validity and competency development during training. Surg Endosc. 2020 Jan;34(1):115. doi: 10.1007/s00464-019-06776-0. PMID 30937617
- [Background] ASGE Training Committee; Sedlack RE, Coyle WJ, Obstein KL, Al-Haddad MA, Bakis G, Christie JA, Davila RE, DeGregorio B, DiMaio CJ, Enestvedt BK, Jorgensen J, Mullady DK, Rajan L. ASGE's assessment of competency in endoscopy evaluation tools for colonoscopy and EGD. Gastrointest Endosc. 2014 Jan;79(1):1-7. doi: 10.1016/j.gie.2013.10.003. Epub 2013 Nov 14. No abstract available. PMID 24239255
- [Background] van Dongen KW, Verleisdonk EJ, Schijven MP, Broeders IA. Will the Playstation generation become better endoscopic surgeons? Surg Endosc. 2011 Jul;25(7):2275-80. doi: 10.1007/s00464-010-1548-2. Epub 2011 Mar 17. PMID 21416186
- [Background] Scaffidi MA, Grover SC, Carnahan H, Yu JJ, Yong E, Nguyen GC, Ling SC, Khanna N, Walsh CM. A prospective comparison of live and video-based assessments of colonoscopy performance. Gastrointest Endosc. 2018 Mar;87(3):766-775. doi: 10.1016/j.gie.2017.08.020. Epub 2017 Aug 30. PMID 28859953
- [Background] Sewell JL, Boscardin CK, Young JQ, Ten Cate O, O'Sullivan PS. Measuring cognitive load during procedural skills training with colonoscopy as an exemplar. Med Educ. 2016 Jun;50(6):682-92. doi: 10.1111/medu.12965. PMID 27170086
- [Background] Sewell JL, Boscardin CK, Young JQ, Ten Cate O, O'Sullivan PS. Learner, Patient, and Supervisor Features Are Associated With Different Types of Cognitive Load During Procedural Skills Training: Implications for Teaching and Instructional Design. Acad Med. 2017 Nov;92(11):1622-1631. doi: 10.1097/ACM.0000000000001690. PMID 28445213
- [Background] Thomas-Gibson S, Saunders BP. Development and validation of a multiple-choice question paper in basic colonoscopy. Endoscopy. 2005 Sep;37(9):821-6. doi: 10.1055/s-2005-870202. PMID 16116532
- [Background] Bini EJ, Firoozi B, Choung RJ, Ali EM, Osman M, Weinshel EH. Systematic evaluation of complications related to endoscopy in a training setting: A prospective 30-day outcomes study. Gastrointest Endosc. 2003 Jan;57(1):8-16. doi: 10.1067/mge.2003.15. PMID 12518123
- [Background] Fudman DI, Falchuk KR, Feuerstein JD. Complication rates of trainee- versus attending-performed upper gastrointestinal endoscopy. Ann Gastroenterol. 2019 May-Jun;32(3):273-277. doi: 10.20524/aog.2019.0372. Epub 2019 Mar 28. PMID 31040624
- See also: certification of endoscopic training by DGVS — http://www.dgvs.de/fortbildung-aktuell/zertifizierung-endoskopischer-trainingskurse/